CLINICAL TRIAL: NCT04811027
Title: TACTI-003 (Two ACTive Immunotherapeutics): A Multicenter, Open Label, Randomized, Phase II Trial to Investigate a Soluble LAG-3 Fusion Protein, Eftilagimod Alpha (Efti; IMP321) in Combination With Pembrolizumab (PD-1 Antagonist) for First Line Treatment of Subjects With Unresectable Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Combination Study With Eftilagimod Alpha (a Soluble LAG-3 Fusion Protein) and Pembrolizumab in Patients With Recurrent or Metastatic HNSCC
Acronym: TACTI-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTI-003; 2021-000055-39 (EudraCT Number); KEYNOTE-C34 (Other: Merck Sharp & Dohme LLC); MK-3475-C34 (Other: Merck Sharp & Dohme LLC); 2024-510762-16-00 (Other: EU CT number)
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: HNSCC
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — soluble LAG-3 protein, human; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- (CPS ≥1): pembrolizumab (KEYTRUDA®) + efti (Experimental): eftilagimod alpha: 30 mg every 2 weeks for the first 4 cycles;thereafter every 3 weeks for up to 18 cycles (1 cycle = 6 weeks).
  pembrolizumab (KEYTRUDA®): 400 mg every 6 weeks for up to 18 cycles (1 cycle = 6 weeks).
  Interventions: Drug: eftilagimod alpha; Drug: pembrolizumab (KEYTRUDA®)
- (CPS ≥1): pembrolizumab (KEYTRUDA®) (Active Comparator): pembrolizumab (KEYTRUDA®): 400 mg every 6 weeks for up to 18 cycles (1 cycle = 6 weeks).
  Interventions: Drug: pembrolizumab (KEYTRUDA®)
- (CPS <1): pembrolizumab (KEYTRUDA®) + efti (Experimental): eftilagimod alpha: 30 mg every 2 weeks for the first 4 cycles;thereafter every 3 weeks for up to 18 cycles (1 cycle = 6 weeks).
  pembrolizumab (KEYTRUDA®): 400 mg every 6 weeks for up to 18 cycles (1 cycle = 6 weeks).
  Interventions: Drug: eftilagimod alpha; Drug: pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: eftilagimod alpha — APC activator, MHC II agonist, LAG-3 fusion protein
  Other Names: IMP321; efti; eftilagimod alfa
  Arms: (CPS <1): pembrolizumab (KEYTRUDA®) + efti; (CPS ≥1): pembrolizumab (KEYTRUDA®) + efti
Drug: pembrolizumab (KEYTRUDA®) — anti-PD-1 antibody
  Other Names: MK-3475

SUMMARY:
Evaluate the safety and efficacy of eftilagimod alpha in combination with pembrolizumab against pembrolizumab alone in 1st line metastatic or recurrent HNSCC with programmed death-ligand 1 (PD-L1) positive (combined positive score [CPS] ≥1) tumors, and determine the efficacy and safety of efti plus pembrolizumab in patients with PD-L1 negative tumors.

DETAILED DESCRIPTION:
Up to 154 patients will be recruited in the TACTI-003 (Two ACTive Immunotherapies) Phase IIb study which will take place across several countries in Australia, Europe and United States of America in up to 35 experienced clinical sites. It will evaluate the safety and efficacy of eftilagimod alpha in combination with pembrolizumab against pembrolizumab alone in 1st line metastatic or recurrent HNSCC with PD-L1 positive (CPS ≥1) tumors, and determine the efficacy and safety of efti plus pembrolizumab in patients with PD-L1 negative tumors. Subjects in cohort A (CPS ≥1) will be randomized 1:1 to receive either "P+E": efti plus pembrolizumab or "P only": pembrolizumab alone. Subjects in cohort B (CPS <1) will receive a combination of efti and pembrolizumab "P+E". Efti will be administered for up to 24 months using a 30 mg subcutaneous dosing every 2 or 3 weeks. Pembrolizumab will be administered for up to 24 months using a 400 mg intravenous (30 min) dosing every 6 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

1. Histologically- or cytologically-confirmed recurrent disease not amenable to curative treatment with local or systemic therapy, or metastatic (disseminated) HNSCC of the oral cavity, oropharynx, hypopharynx, or larynx that is considered incurable by local therapies and to be treated in the first line palliative setting and who are PD-X naïve.
2. Availability of tissue for PD-L1 biomarker analysis from a core or excisional biopsy.
3. Availability of PD-L1 biomarker result by using the FDA approved Dako standardized diagnostic test (PD-L1 IHC 22C3 pharmDx).
4. Availability of tissue for testing of human papillomavirus (HPV) status for oropharyngeal cancer (p16 expression testing).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Main Exclusion Criteria:

1. Disease is suitable for local therapy administered with curative intent.
2. Previously treated with ≥ 1 systemic regimen for recurrent and/or metastatic disease (with the exception of systemic therapy completed >6 months prior if given as part of multimodal treatment for locally or locoregionally advanced disease).
3. Histologically or cytologically confirmed head and neck cancer of any other primary anatomic location in the head and neck not specified in the inclusion criteria including subjects with HNSCC of unknown primary, squamous cell carcinoma originating from skin, or non-squamous histologies (e.g. nasopharynx, salivary gland or mucosal melanoma).
4. Has progressive disease (PD) within 6 months of completion of curatively intended systemic treatment for locally or locoregionally advanced HNSCC, or requires chemotherapy based therapeutic regimen due to e.g., rapidly progressing disease or need of aggressive sympton control.
5. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
6. Has received prior chemotherapy, anti-cancer monoclonal antibody, major surgery, another systemic cancer therapy or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to cycle 1 day 1.
7. Known active central nervous system metastasis and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable: i.e. without evidence of progression documented by repeat imaging performed after therapy completed for CNS metastasis and with at least 4 weeks difference, clinically stable and without requirement for steroid treatment for at least 14 days prior to cycle 1 day 1.
8. Receives continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days prior to cycle 1 day 1. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalents are permitted in the absence of active auto-immune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 24 months

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
Objective response rate (ORR) according to iRECIST | Up to 24 months
Duration of responses according to iRECIST and RECIST 1.1 | Up to 24 months
Disease control rate according to iRECIST and RECIST 1.1 | Up to 24 months
Progression free survival (PFS) according to iRECIST and RECIST 1.1 | Up to 24 months
Frequency of (serious) adverse events | Up to 24 months
Severity of (serious) adverse events according to the United States National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v5.0 | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (28):
- United States (3):
  - University of Alabama at Birmingham (UAB) - O'Neal Cancer Center, Birmingham, Alabama
  - Washington University School of Medicine, St Louis, Missouri
  - Oncology Consultants, Houston, Texas
- Macquarie University Hospital, Macquarie Park, New South Wales, Australia
- Belgium (4):
  - AZ Sint-Jan Brugge, Bruges
  - Antwerp University Hospital, Edegem
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
  - AZ Nikolaas, Sint-Niklaas
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
- Germany (4):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Essen, Essen
  - Nationales Centrum für Tumorerkrankungen Heidelberg, Heidelberg
  - Universitätsklinikum Ulm, Ulm
- The Oncology Institute "Prof Dr Ion Chiricuta" I.O.C.N., Cluj-Napoca, Romania
- Spain (8):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Institut Català d'Oncologia - Hospital Universitari de Girona, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - START Madrid (Hospital Universitario Fundación Jiménez Díaz), Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Arensia Exploratory Medicine Llc, Kapitanivka, AL, Ukraine
- United Kingdom (4):
  - Institute of Cancer Science - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospitals NHS Foundation - The Harley Street Clinic, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals, NHS Trust, Nottingham